CLINICAL TRIAL: NCT05812521
Title: Efficacy of Thoracic Paravertebral Block With Methylene Blue Visual Confirmation in the Management of Postoperative Pain After Video-assisted Thoracoscopic Lobectomy
Brief Title: Thoracic Paravertebral Block With Methylene Blue Visual Confirmation for Postoperative Pain After VATS Lobectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Alfonso Fiorelli, Full Professor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29917/2022
Record Dates: First submitted 2023-03-19; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Post Operative Pain; Thoracic Cancer
Keywords: postoperative pain; regional anesthesia; thoracoscopy
MeSH Terms: conditions — Pain, Postoperative | interventions — Methylene Blue

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paravertebral block with methylene blue (Experimental): With the patient sitting, the patient will receive paravertebral block at T4-T5 level before general anesthesia induction
  Interventions: Procedure: Paravertebral block with methylene blue
- Thoracic Epidural Anesthesia (Active Comparator): With the patient sitting, the patient will receive thoracic epidural anesthesia at T4-T8 level before general anesthesia induction
  Interventions: Procedure: Thoracic Epidural Anesthesia

INTERVENTIONS:
Procedure: Paravertebral block with methylene blue — The paravertebral space is identified under ultrasound guidance and after negative aspiration a 3 ml test dose of anesthetic is injected. After observing widening of the paravertebral space and anterior pleural displacement to confirm the correct needle positioning, a bolus dose of 20 mL 0.5% ropivacaine with a solution of 1 ml 1% methylene blue and 4 ml of saline will be injected in the paravertebral space. At the start of the surgery, the spread of the solution of anesthetic and methylene blue will be assessed through visualization in thoracoscopy and if necessary the block will be repeated. After the surgery, intravenous acetaminophen will be administered 3 times daily and tramadol 50 mg will be prescribed as rescue analgesic.
  Arms: Paravertebral block with methylene blue
Procedure: Thoracic Epidural Anesthesia — The epidural catheter will be placed using the loss of resistance technique, and after ruling out intravenous or intrathecal catheter placement with a negative aspiration test dose, an initial dose of 10 mL 0.25% bupivacaine will be injected. Continuous infusion will be started with with 0.125 % bupivacaine + fentanyl 0.5 mcg/ ml at 6-10 ml/hour will be started based on the patient weight for 48 hours postoperatively. After the surgery, intravenous acetaminophen will be administered 3 times daily and tramadol 50 mg will be prescribed as rescue analgesic.
  Arms: Thoracic Epidural Anesthesia

SUMMARY:
The goal of this study is to compare the efficacy in controlling postoperative pain of paravertebral block (PVB) with methylene blue visual confirmation and thoracic epidural anesthesia (TEA). This is a single center, parallel-group, prospective study. Patients will be randomly assigned in a 1:1 ratio to receive either PVB or TEA. Primary end-point is pain relief measured with Postoperative Numeric Rating Scale. The secondary end-points are time to perform TEA and PVB, total opioid consumption, postoperative outcomes.

DETAILED DESCRIPTION:
The management of postoperative pain in patients undergoing thoracoscopic lobectomy is a fundamental part of the process of recovery. Uncontrolled thoracic pain in the early postoperative period may interfere with the mobilization of the patients, leading to increased morbidity and reduction in the quality of life.

Thoracic paravertebral block (PVB) is an effective strategy for controlling postoperative pain after video-assisted thoracoscopic (VATS) lobectomy, but it may be subjected to a high rate of failure due to incorrect identification of the site of local anesthetic injection.

Thoracic epidural anesthesia (TEA) is considered a reliable technique for regional thoracic anesthesia, however potential side effects may limit its use.

Herein the investigators reported a new technique using methylene blue as a visual confirmation of the correct anesthetic diffusion during PVB. Then, the investigators will compare the efficacy of methylene blue PVB with TEA for the management of postoperative pain in patients undergoing VATS lobectomy.

This is a single center, parallel-group, prospective study. Participants will be randomly assigned in a 1:1 ratio to receive either PVB with methylene blue or TEA.

All participants will receive postoperatively intravenous acetaminophen as additional analgesics and intravenous tramadol as rescue analgesic. Primary end-point is pain relief measured with Postoperative Numeric Rating Scale at at 1, 12, 24, 48 hours postoperatively. The secondary end-points are: (i) time to perform TEA and PVB, (ii) total opioid consumption, (iii) postoperative outcomes (including complications, chest drainage duration and length of hospital stay).

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 - 85 years old
* scheduled to undergo thoracoscopic lobectomy for lung cancer
* standardized three-port anterior thoracoscopic approach

Exclusion Criteria:

* Allergy to any of the drugs used in the study
* Previous thoracic surgical procedures or lung resection
* Psychiatric disorders
* ASA (American Society of Anesthesiologists) Class > III
* Conversion to thoracotomy
* Lack of written informed consent
* Participation to other studies
* Contraindications to epidural analgesia or paravertebral block

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Pain Scores on the Postoperative Numeric Rating Scale in the first 48 hours postoperatively | 1 hours, 12 hours, 24 hours and 48 hours after surgery
  Pain scores at rest and after cough will be evaluated in the first 48 hours postoperatively using Postoperative Numeric Rating Scale (NRS) ranging from 0 (absence of pain) to 10 (maximum level of pain)

SECONDARY OUTCOMES:
Opioids consumption | through the entire hospital stay, an average of 8 days"
  Cumulative dose of intravenous opioids administered as rescue analgesic will be registered during the post-operative period.
Time to perform PVB or TEA | From the identification of the site of injection to the start of general anesthesia, up to 1 hour
  Time needed to perform PVB or TEA will be recorded
Chest tube duration | From chest tube placement to chest tube removal, up to 20 days
  Total days of chest tube duration will be recorded
Length of hospital stay | From hospital admission to discharge, up to 20 days
  Total days of hospital stay will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Fiorelli, MD, PhD, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Alfonso Fiorelli, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yeap YL, Wolfe JW, Backfish-White KM, Young JV, Stewart J, Ceppa DP, Moser EAS, Birdas TJ. Randomized Prospective Study Evaluating Single-Injection Paravertebral Block, Paravertebral Catheter, and Thoracic Epidural Catheter for Postoperative Regional Analgesia After Video-Assisted Thoracoscopic Surgery. J Cardiothorac Vasc Anesth. 2020 Jul;34(7):1870-1876. doi: 10.1053/j.jvca.2020.01.036. Epub 2020 Jan 25. PMID 32144059
- [Background] D'Ercole F, Arora H, Kumar PA. Paravertebral Block for Thoracic Surgery. J Cardiothorac Vasc Anesth. 2018 Apr;32(2):915-927. doi: 10.1053/j.jvca.2017.10.003. Epub 2017 Oct 4. PMID 29169795
- [Background] Norum HM, Breivik H. A systematic review of comparative studies indicates that paravertebral block is neither superior nor safer than epidural analgesia for pain after thoracotomy. Scand J Pain. 2010 Jan 1;1(1):12-23. doi: 10.1016/j.sjpain.2009.10.003. PMID 29913936
- [Background] Baidya DK, Khanna P, Maitra S. Analgesic efficacy and safety of thoracic paravertebral and epidural analgesia for thoracic surgery: a systematic review and meta-analysis. Interact Cardiovasc Thorac Surg. 2014 May;18(5):626-35. doi: 10.1093/icvts/ivt551. Epub 2014 Jan 31. PMID 24488821
- [Background] Casati A, Alessandrini P, Nuzzi M, Tosi M, Iotti E, Ampollini L, Bobbio A, Rossini E, Fanelli G. A prospective, randomized, blinded comparison between continuous thoracic paravertebral and epidural infusion of 0.2% ropivacaine after lung resection surgery. Eur J Anaesthesiol. 2006 Dec;23(12):999-1004. doi: 10.1017/S0265021506001104. Epub 2006 Jul 7. PMID 16824243
- [Background] Helms O, Mariano J, Hentz JG, Santelmo N, Falcoz PE, Massard G, Steib A. Intra-operative paravertebral block for postoperative analgesia in thoracotomy patients: a randomized, double-blind, placebo-controlled study. Eur J Cardiothorac Surg. 2011 Oct;40(4):902-6. doi: 10.1016/j.ejcts.2011.01.067. Epub 2011 Mar 5. PMID 21377888
- [Background] Ding X, Jin S, Niu X, Ren H, Fu S, Li Q. A comparison of the analgesia efficacy and side effects of paravertebral compared with epidural blockade for thoracotomy: an updated meta-analysis. PLoS One. 2014 May 5;9(5):e96233. doi: 10.1371/journal.pone.0096233. eCollection 2014. PMID 24797238
- [Background] Marshall K, McLaughlin K. Pain Management in Thoracic Surgery. Thorac Surg Clin. 2020 Aug;30(3):339-346. doi: 10.1016/j.thorsurg.2020.03.001. Epub 2020 Apr 29. PMID 32593366